CLINICAL TRIAL: NCT01802736
Title: Alcohol Consumption and Alcohol Reduction Intervention Among HIV Infected Persons in a Large Urban HIV Clinic in Uganda
Brief Title: Alcohol Use and Risky Sexual Behaviors Among HIV Infected Subjects in Kampala Uganda
Acronym: ASK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Training Health research into Vocational excellence in East Africa (THRiVE) (Unknown); Wellcome Trust (Other); Infectious Diseases Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THRiVE- ASK
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Alcohol Use; HIV
Keywords: Alcohol HIV intervention counselling; Alcohol Use in HIV infected Persons
MeSH Terms: conditions — Alcohol Drinking | interventions — signal peptide peptidase; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Positive Prevention Counselling (Active Comparator): Standard positive prevention counseling which includes alcohol reduction and sexual risk behavior counseling provided in the clinic by the clinic medical counselors on the day of enrollment and at month 3 visit.
  Although there is awareness of the need to engage and include PLWHA in HIV prevention, there are little practical efforts devoted towards this engagement even in developed countries. One of the major reasons is the lack of a well-defined standard positive prevention package that needs to be delivered to PLWHA. The approach proposed by Kennedy et al modified to suit the local setting and involves a simpler understandable classification of the goals, interventions and expected outcomes of the treatment.
  Interventions: Behavioral: Motivational intervention counselling plus SPP
- Alcohol Motivational intervention counselling plus SPP (Experimental)
  Interventions: Behavioral: Motivational intervention counselling plus SPP

INTERVENTIONS:
Behavioral: Motivational intervention counselling plus SPP
  Other Names: Alcohol Motivational Intervention counseling plus Standard Positive Prevention Counselling

SUMMARY:
Background: Approximately 6.4% of Ugandans are living with HIV, that is acquired and transmitted mainly through sexual intercourse between an HIV infected and uninfected person. Uganda is ranked among 28 top per capita alcohol consumers in the world and second in Africa. in the general population, Alcohol consumption is associated with increased sexual transmission risks for HIV. Data on alcohol consumption and its impact on sexual behaviors and HIV disease progression among HIV infected persons, the persons able to transmit HIV are lacking in this setting.

Objectives: To estimate the prevalence of alcohol consumption among HIV infected persons, assess associations between alcohol and CD4 cell count as well as evaluate the effect of alcohol motivational intervention counseling on alcohol consumption and the subsequent practice of risky sexual behaviors, among HIV infected persons.

Methodology: Using both cross-sectional and longitudinal methods,persons living with HIV/AIDS (PLWHA) attending the Infectious Diseases Institute Clinic (IDI clinic) will be recruited, baseline alcohol consumption evaluated, and eligible subjects reporting alcohol consumption will be randomized to receive either Standard positive prevention counseling alone or in addition to alcohol motivation intervention counseling. Sexual risk behaviors and alcohol consumption will be evaluated at 3 and 6 months and compared between randomization arms.

DETAILED DESCRIPTION:
Uganda is among countries with the highest per capita consumption rates of alcohol as well as a high prevalence of HIV. Uganda is ranked the 28th in the world in alcohol consumption per capita and is 2nd top consumer of alcohol in Africa.

Little is known about alcohol use and its impact on sexual risk behaviors and HIV disease progression from this setting Understanding alcohol consumption burden and testing an intervention measure directed against alcohol consumption will result in reduced alcohol consumption and potentially reduced sexual risk behaviors hence boost the success of ART and subsequently reduce potential further HIV transmission from Persons Living With HIV/AIDS.

To increase the understanding of alcohol consumption among persons living with HIV in through a series of epidemiological studies by estimating the burden of alcohol consumption, its association with HIV disease progression and assess the effect of an alcohol motivational intervention plus standard positive prevention versus standard positive prevention counseling alone on alcohol and sexual risk behaviors among PLWHA at the IDI clinic.

Specific Objectives

1. To identify and determine the prevalence of clinical factors associated with any alcohol consumption among PLWHA attending the IDI clinic in Kampala Uganda
2. To describe the association between moderate alcohol consumption and CD4 cell count at base-line among patients attending the IDI clinic.
3. To determine the efficacy of standard positive prevention counseling plus Motivational intervention (SPP+MI) for alcohol consumption versus standard positive prevention counseling (SPP) only in reducing alcohol consumption among HIV infected moderate alcohol drinkers attending the IDI clinic in Kampala Uganda.
4. To determine whether reduction in alcohol consumption is associated with reductions in risky sexual behaviors among HIV infected moderate alcohol drinkers attending the AIDC in Kampala Uganda.

Risky Sexual Behavior for HIV transmission assessed as a summation of yes or no(Binary) if reporting ANY ONE or ALL of the following behaviors (non spousal sexual inter-course, unprotected sex with any partner who is HIV negative/unknown HIV status or reporting multiple Non spousal sex partners within the study period under inquiry.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females aged at least 18 years.
* Willing to continue receiving care /be followed up at the IDI for the next 6 months.
* Willing to provide written informed consent.

Exclusion Criteria:

* Very sick with Karnofsky clinical performance score < 50.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol consumption Score as assessed by the AUDIT-C tool . | 6 months

SECONDARY OUTCOMES:
Change in Risky sexual behavior composite in the last 3 months assessed at baseline, 3 and 6 month visit. | 3 and 6 months

OTHER OUTCOMES:
CD4 Cell count in the last 6 months preceding the study visit | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

REFERENCES:
- [Derived] Greene MC, Kane J, Alto M, Giusto A, Lovero K, Stockton M, McClendon J, Nicholson T, Wainberg ML, Johnson RM, Tol WA. Psychosocial and pharmacologic interventions to reduce harmful alcohol use in low- and middle-income countries. Cochrane Database Syst Rev. 2023 May 9;5(5):CD013350. doi: 10.1002/14651858.CD013350.pub2. PMID 37158538
- [Derived] Wandera B, Tumwesigye NM, Nankabirwa JI, Mafigiri DK, Parkes-Ratanshi RM, Kapiga S, Hahn J, Sethi AK. Efficacy of a Single, Brief Alcohol Reduction Intervention among Men and Women Living with HIV/AIDS and Using Alcohol in Kampala, Uganda: A Randomized Trial. J Int Assoc Provid AIDS Care. 2017 May/Jun;16(3):276-285. doi: 10.1177/2325957416649669. Epub 2016 May 23. PMID 27215561